CLINICAL TRIAL: NCT02922595
Title: Comparison of iLTS-D® and ILMA® for Intubation With Fiberoptic Control. Multicentric Randomised Patient-blind Study of Non-inferiority
Brief Title: Comparison of iLTS-D® and ILMA® for Intubation With Fiberoptic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patrick Schoettker,MD PD (Other)
Responsible Party: Sponsor-Investigator, Patrick Schoettker,MD PD, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-00902
Record Dates: First submitted 2016-09-21; First posted 2016-10-04 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intubation through ILMA® (Active Comparator): The ILMA will be placed into patient's larynx through the mouth in accordance with manufacturer's recommendations by experienced airway providers. The Intervention will be the intubation through ILMA. We will measure the time necessary to insert it, the possibility to ventilate the patient through it and the success rate of tracheal intubation through it will be assessed.
  Interventions: Device: Intubation through ILMA®
- Intubation through ILTS® (Experimental): The ILTA will be placed into patient's larynx through the mouth in accordance with manufacturer's recommendations by experienced airway providers. It will be proceeded to the intubation through ILTS and the time necessary to insert it, the possibility to ventilate the patient through it and the success rate of tracheal intubation through it will be assessed.
  Interventions: Device: Intubation through ILTS®

INTERVENTIONS:
Device: Intubation through ILMA® — It will be placed into patient's larynx through the mouth in accordance with manufacturer's recommendations by experienced airway providers.
  Intubation will then be peformed
  Arms: Intubation through ILMA®
Device: Intubation through ILTS® — It will be placed into patient's larynx through the mouth in accordance with manufacturer's recommendations by experienced airway providers.
  Intubation will then be peformed
  Arms: Intubation through ILTS®

SUMMARY:
The primary purpose of this study is to compare with a non-inferiority randomised study the new laryngeal tube (Intubating Laryngeal Tube Single-Disposable - iLTS-D) to the well-established Intubating Larygeal Mask Airway (ILMA/ Fastrach) for the success rate and time for intubation under fiberoptic control. Secondary purposes are success rates and times for ventilation for both devices and finally success rate of gastric tube placement.

DETAILED DESCRIPTION:
During general anesthesia or for some life-threatening conditions (unconsciousness, respiratory insufficiency), tracheal intubation may be mandatory. Tracheal intubation consists of inserting a tube inside the trachea through the glottis, therefore allowing patients' ventilation and airway protection. However, in some cases, intubation can be difficult with standard method (e.g. direct laryngoscopy) and visualisation of the glottis may be impossible. In those cases, alternative devices may be successful (e.g. videolaryngoscopy, fiberscopy). In cases of failure of alternative devices, prioritization to patients' ventilation is mandatory and supra-glottic devices like laryngeal masks and tubes are designed to allow an adequate ventilation. These devices are present in all difficult intubations algorithms and represent a mandatory alternative. For some specific models, tracheal intubation is possible through some of the supra-glottic devices. It's the case for the ILMA, which remains, despite the fact being more than 20 years old, the Gold Standard. Until now, no other supra-glottic device equals the ILMA concerning blind intubation, which is often necessary in emergency situations or outside the operating room (e.g. out-of-hospital care).

The design and 2016 market release of a new laryngeal tube which equally allows intubation through the device (iLTS-D) and has a gastric access potentially challenges the supremacy of the ILMA. The first two studies concerning the iLTS-D have shown encouraging results. A first study made on manikins showed a similar success rate and time for intubation for the ILMA and iLTS-D, while the insertion of the LTS-D being easier and quicker than the ILMA. A second one has demonstrated a success intubation through the iLTS-D in 29 patients of 30 without any difficult intubation criteria with 2 attempts under fiberoptic control. Concerning ventilation, the iLTS-D doesn't differ of the already well-known LTS-D.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Adult patients who will undergo an elective surgery under general anesthesia requiring tracheal intubation
* American Society of Anesthesiology ASA Risk Class 1-3

Exclusion Criteria:

* Known difficult intubation
* Previous surgery of Ear Nose Throat (ENT)
* Symptomatic gastrooesophageal reflux
* Nauseas at time of operation
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
success rate intubation | 60 minutes
  The primary endpoint will be the success rate for tracheal intubation under fiberoptic control through both devices. Intubation for patients with difficult airways is the main feature of those devices.
time necessary to intubate | 180 seconds
  We will measure the time necessary to intubate

SECONDARY OUTCOMES:
success rate ventilation | 60 minutes
  Secondary endpoint will be success rate for ventilation for both devices
time to ventilation | 180 seconds
  Secondary endpoint will be time necessary to achieve for ventilation for both devices
time to intubation | 180 seconds
  Secondary endpoint will be time necessary for intubation for both devices

CONTACTS AND LOCATIONS:
Overall Officials: patrick Schoettker, Professor, Study Director — University Hospital Lausanne CHUV
Locations (1):
- Dpt of Anesthesiology, University of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuercher M, Casso G, Krugel V, Potie A, Barry MP, Schoettker P. Tracheal intubation using intubating laryngeal tube iLTS-D and LMA Fastrach in 99 adult patients: A prospective multicentric randomised non-inferiority study. J Clin Anesth. 2022 Jun;78:110671. doi: 10.1016/j.jclinane.2022.110671. Epub 2022 Feb 9. PMID 35151143